CLINICAL TRIAL: NCT04877535
Title: A Pilot Study for the Effect of Risk Prediction on Anticipatory Guidance and Team Coordination for Postoperative Care
Brief Title: Pilot Study for Postoperative Machine Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202103210; KL2TR002346 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Surgery--Complications
Keywords: Telemedicine; Anesthesia Control Tower; Machine Learning; Forecasting Algorithms; Handoff effectiveness

STUDY DESIGN:
Intervention Model Description: Blended pre-post and parallel design. Participants will be allocated to up to two groups in two time periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Stage 2: Intervention (Experimental): ML will be used to create a report card for each patient that summarizes the preoperative assessment and intraoperative data. Report card data will be made available to providers through multiple methods: integration into electronic health records workflows, electronic health records notifications, mobile device notifications, and print outs in the paper chart
  Patients who have a previous assignment (from another day) are not eligible.
  Interventions: Device: ML-based report card
- Stage 2: Usual Care (No Intervention): The standard of care. The report card will be electronically generated (to determine eligibility) but it will not be visible to clinicians.
  Patients who have a previous assignment (from another day) are not eligible.
- Stage 1: Usual Care (No Intervention): The standard of care. The report card will be electronically generated (to determine eligibility) but it will not be visible to clinicians.

INTERVENTIONS:
Device: ML-based report card — PACU and ward providers caring for participants will be notified by Anesthesia Control Tower clinicians before arrival if the patient's report card. The notification will contain a report card of the patient's forecast risk of major adverse events, explanatory machine-learning outputs, most influential pre- and intraoperative data, and predicted treatments.The ML risk profile generated for each patient will include risk of 30 day mortality, risk of respiratory failure, risk of acute kidney injury, and risk of postoperative delirium
  Arms: Stage 2: Intervention

SUMMARY:
The objectives of the study are to determine the interpretability, workflow role, and effect on communications of showing report cards containing Machine Learning (ML)-based risk profiles based on pre- and intra-operative data to postoperative providers.

DETAILED DESCRIPTION:
Although surgery and anesthesia have become much safer on average, many patients still experience complications after surgery. Some of these complications are likely to be avoided or less severe with early detection and treatment. Barnes-Jewish Hospital has recently started using an Anesthesia Control Tower (ACT), which is a remote group lead by an anesthesiologist who reviews live data from BJH operating rooms and calls the anesthesia provider with concerns to improve reaction times and improve use of best-practices treatments. The ACT also uses machine learning (ML) to calculate patient risks during surgery as a way of measuring when the patient is doing better or worse.

The study team suspects that two mechanisms may allow risk prediction to improve postoperative care. First, is that it may make some data more actionable to clinicians. Although intraoperative data is extremely rich with many monitors, drug-response events, and surgical stress reactions to reveal the physiological state of the patient, that data is also extremely specialized and difficult to access. The study team thinks that many times the right interpretation of intraoperative data or the right treatment to give isn't clear until the surgery is nearly finished. The medical team in the recovery room (post-anesthesia care unit, PACU) and surgical wards is responsible for deciding the treatment strategy, but they don't have access to the information from the intraoperative monitors and events. Those providers also lack the familiarity to directly interpret that information and time to review it in detail. Even preoperative information may be less than fully available because the patient may still be too sedated or confused from the anesthesia to explain much about their history. By summarizing these diverse sources of information into a risk profile, machine learning outputs may directly improve the understanding of postoperative providers or improve the identification of patients at elevated risk for postoperative adverse outcomes.

A second mechanism derives from behavior changes which may occur in providers in reaction to machine-generated risk profiles. The study team has observed many handoffs from the operating room and PACU include lists of "important" data, but it is common for the handoff-giver to provide no interpretation (what problem is this information related to) or anticipatory guidance (having identified a potential or actual problem, what should the handoff receiver do). The study team has also observed than once a major risk has been clearly identified along the chain of handoff it tends to be propagated forward with connection to the underlying data, any changes noticed by the current provider, and the current plan. The study team suspects that in the subset of patients with substantially elevated predictions on their risk profile, handoff communication and team coordination for the identified problems may improve.

The larger goal is to deploy a "report card" for each patient that summarizes the preoperative assessment and intraoperative data in a way that is useful for postoperative providers. In this study these ML reports will be integrated into the clinical workflow and determine if it does affect handoff behavior. The study team will also evaluate the information-effect and test the report card for safety by determining if clinicians identify any major inaccuracies related to the implementation.

This study is a substudy of a randomized trial of ACT-intraoperative contact (TECTONICS IRB# 201903026), and only patients in the contact (treatment) group will be eligible. The screened patients will be all adults having surgery at BJH with the division of Acute and Critical Care Surgery. Exclusion criteria are a planned ICU admission. For each included patient, the ACT clinician will review the report card information, and the postoperative providers will either be directly contacted or receive an Epic Best Practices Advisory. Our study will be a before-after quasi-experiment, meaning that after a fixed date, all eligible patients will receive the intervention, and the outcome measures will be compared to patients before that date. The outcome measure we will study is handoff effectiveness from the recovery room to wards. Providers will be surveyed on information value, any inaccurate items, or major omissions.

The ML report card will not recommend specific treatments, and decisions will remain the hands of the physician in the PACU or wards. The postoperative provider will also be given information about the report card and its limitations.

Modifications during piloting We originally intended the report data to be included in the electronic medical record hand off workflow for the pacu receiving nurse, however, due to changes in institutional priorities this was not activated.

The study was originally designed as a pre- versus post-intervention comparison. However, it was apparent during pre-intervention data collection (June 3 2021 - July 22 2021) that differences in individual research-assistant's evaluation of hand-off content and changes in other behavior would make this a low validity method. After 2 months, the design was changed to a non-randomized parallel group study with alternating days with the report card turned on or off in a 2:1 ratio. We also took this opportunity to expand the inclusion criteria to include patients with vascular surgery, as they were frequently identified as high-risk.

Due to a lack of staff availability, no further enrollment was attempted until October 2022. Enrollment continued from Oct 11 2022 to May 11 2023, with no enrollment in Jan or Feb 2023 due to staff availability.

ELIGIBILITY:
Inclusion Criteria:

ODIN-Pilot will intervene on a subset of TECTONICS participants meeting all the following criteria:

1. Within the TECTONICS contact arm (adults undergoing OR procedures)
2. Operating room at BJH South campus (including all of "Pod 2", "Pod 3", "Pod 5") (excluding all procedure suites such as Interventional Radiology, Parkview Tower "Pod 1", Center for Advanced Medicine "Pod 4", Labor and Delivery suites)
3. Surgeon is a member of the Acute and Critical Care Surgery division or the postoperative bed is 16300 observation unit.
4. Planned non-ICU disposition ("floor" and "observation unit" collectively "ward" patients).

Exclusion Criteria:

1. Not enrolled in TECTONICS Study
2. Randomized to the observation arm in TECTONICS study
3. Planned ICU admission
4. Patients are only included once; if previously included a subsequent surgery is not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R King, MD, PhD, Principal Investigator — Washington Univeristy School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data are a subset of TECTONICS and will be have the same sharing plan / restrictions.

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 2: Intervention: ML will be used to create a report card for each patient that summarizes the preoperative assessment and intraoperative data. Report card data will be made available to providers through multiple methods: integration into electronic health records workflows, electronic health records notifications, mobile device notifications, and print outs in the paper chart
  ML-based report card: PACU and ward providers caring for participants will be notified by Anesthesia Control Tower clinicians before arrival if the patient's report card. The notification will contain a report card of the patient's forecast risk of major adverse events, explanatory machine-learning outputs, most influential pre- and intraoperative data, and predicted treatments.The ML risk profile generated for each patient will include risk of 30 day mortality, risk of respiratory failure, risk of acute kidney injury, and risk of postoperative delirium
  Patients who have a previous assignment (from another day) are not eligible.
Period: Overall Study
Arm/Group | Stage 1: Usual Care | Stage 2: Usual Care | Stage 2: Intervention
Started | 89 | 39 | 94
Completed | 89 | 39 | 94
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants analyzed
Groups:
- Stage 1: Usual Care: Pre-intervention period
- Stage 2: Usual Care: Days with ML report card disabled
- Stage 2: Intervention: Days with ML report card enabled
- Total: Total of all reporting groups
Arm/Group | Stage 1: Usual Care | Stage 2: Usual Care | Stage 2: Intervention | Total
Number analyzed (Participants) | 89 | 39 | 94 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (15.5) | 62.5 (16.7) | 57.3 (16.5) | 57.9 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 16 | 36 | 98
  Male | 43 | 23 | 58 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 85 | 37 | 92 | 214
  Unknown or Not Reported | 2 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 12 | 31 | 60
  White | 69 | 25 | 59 | 153
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Surgery type [Count of Participants; unit: Participants]
  Acute Critical Care Surgery | 28 | 4 | 13 | 45
  Orthopaedics | 2 | 13 | 40 | 55
  Otolaryngology | 12 | 6 | 11 | 29
  Plastics | 4 | 8 | 4 | 16
  Transplant | 30 | 1 | 2 | 33
  Vascular | 0 | 7 | 22 | 29
  Hepatobiliary | 11 | 0 | 2 | 13
  Unknown or Other | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Handoff Effectiveness
Description: After handoff was completed, receiving nurses were asked:
  Globally, how effective was the handover
  1. Not at all effective
  2. Somewhat effective
  3. Moderately effective
  4. Very effective
  5. Extremely effective
  The item is taken from PMID:25806398 but has no name
Time Frame: 8 hours postop
Measure: Mean (Standard Deviation); unit: score on a 0-5 scale
Arm/Group | Stage 1: Usual Care | Stage 2: Usual Care | Stage 2: Intervention
Number analyzed (Participants) | 89 | 39 | 94
score on a 0-5 scale | 3.9 (0.4) | 3.9 (0.7) | 4.0 (0.7)
Statistical Analysis 1: Comparison: Stage 1: Usual Care vs Stage 2: Intervention; Test type: Superiority; p = 0.524, t-test, 2 sided; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.24 to 0.12]
Statistical Analysis 2: Comparison: Stage 2: Usual Care vs Stage 2: Intervention; Test type: Superiority; p = 0.403, t-test, 2 sided; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.4 to 0.16]

2. Secondary Outcome: Number of Participants With ML Topics Discussed During Handoff
Description: Binary. A research assistant observed the handoff and recorded if any topics identified by the ML algorithm (in the report card) were discussed included in the handoff
Time Frame: 8 hours postop
Population: pre-intervention group did not have ML topics generated for research assistant
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Usual Care | Stage 2: Usual Care | Stage 2: Intervention
Number analyzed (Participants) | 0 | 39 | 94
Participants | 0 | 19 | 47
Statistical Analysis 1: Comparison: Stage 2: Usual Care vs Stage 2: Intervention; Test type: Superiority; p = 1.00, Fisher Exact; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.47 to 2.38]

3. Secondary Outcome: Number of Participants With Anticipatory Guidance During Handoff
Description: Binary. A research assistant observed the handoff and recorded if expected problems or plans to address expected problems were conveyed, or if no expected problems or plans to address expected problems were conveyed.
Time Frame: 8 hours postop
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Usual Care | Stage 2: Usual Care | Stage 2: Intervention
Number analyzed (Participants) | 89 | 39 | 94
Participants | 61 | 35 | 85
Statistical Analysis 1: Comparison: Stage 1: Usual Care vs Stage 2: Intervention; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 4.30, 95% CI 2-sided [1.81 to 11.13]
Statistical Analysis 2: Comparison: Stage 2: Usual Care vs Stage 2: Intervention; Test type: Superiority; p = 1.00, Fisher Exact; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.23 to 4.19]

4. Secondary Outcome: Number of Handoff Receivers Agreeing That They Received All Needed Information
Description: Receiving nurses were asked:
  Did you receive at handoff all the information you needed to safely take care of this patient? [Yes, No]
Time Frame: 8 hours postop
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Usual Care | Stage 2: Usual Care | Stage 2: Intervention
Number analyzed (Participants) | 89 | 39 | 94
Participants | 72 | 37 | 91
Statistical Analysis 1: Comparison: Stage 1: Usual Care vs Stage 2: Intervention; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 7.1, 95% CI 2-sided [1.94 to 39.25]
Statistical Analysis 2: Comparison: Stage 2: Usual Care vs Stage 2: Intervention; Test type: Superiority; p = 0.630, Fisher Exact; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.13 to 14.86]

5. Other Pre Specified Outcome: Number of Handoff Recipients Self-reporting Referring to Report Card OR Report Card Observed Directly Referred to During Handoff
Description: Handoff was observed by a research assistant. In the intervention group only, each nurse was asked
  Did you look at or discuss the postoperative report card for this patient? [Yes, No]
  Additionally, the research assistant noted if they observed the report card being referred to be the handoff-giving team.
  [Yes, No]
  The measure is positive if either the self report or research-assistant recorded a "Yes"
Time Frame: 8 hours postop
Population: Usual care group not eligible
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2: Intervention: ML will be used to create a report card for each patient that summarizes the preoperative assessment and intraoperative data. Report card data will be made available to providers through multiple methods: integration into electronic health records workflows, electronic health records notifications, mobile device notifications, and print outs in the paper chart
  ML-based report card: PACU and ward providers caring for participants will be notified by Anesthesia Control Tower clinicians before arrival if the patient's report card. The notification will contain a report card of the patient's forecast risk of major adverse events, explanatory machine-learning outputs, most influential pre- and intraoperative data, and predicted treatments.The ML risk profile generated for each patient will include risk of 30 day mortality, risk of respiratory failure, risk of acute kidney injury, and risk of postoperative delirium
- Stage 2: Usual Care; Stage 1: Usual Care: The standard of care. The report card will be electronically generated (to determine eligibility) but it will not be visible to clinicians.
  No participants are eligible for this measure.
Arm/Group | Stage 2: Intervention | Stage 2: Usual Care | Stage 1: Usual Care
Number analyzed (Participants) | 94 | 0 | 0
Participants | 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 hours
Groups:
- Stage 2: Intervention Group: Days with ML report card enabled
Arm/Group | Stage 1: Usual Care | Stage 2: Usual Care | Stage 2: Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/39 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/39 | 0/94
Other Adverse Events (participants affected / at risk) | 0/89 | 0/39 | 0/94

LIMITATIONS AND CAVEATS:
During the intervention, we observed that despite education and encouragement, few OR nurses included the report card with the paperwork for the PACU nurse. We determined that the study was unlikely to meet its goals with poor intervention uptake and stopped the trial. In 3 interviews with staff, we found that the workflow was difficult to remember. Because only 2-5 patient per day were eligible, and because of "control" days, staff forget what they were supposed to do with the report card.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT04877535/Prot_SAP_000.pdf